CLINICAL TRIAL: NCT02094859
Title: GlucoClearTM System ICU Study
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Collaborators: MedPass International (Industry); 95 bis boulevard Pereire (Unknown); 75017 Paris - France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012-05
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Accurate Blood Glucose Monitoring in Critical Care Setting
Keywords: Glucose Monitoring

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GlucoClear System

SUMMARY:
The primary purpose of this Study is evaluation of the safety and performance of the GlucoClear System (System).

The primary safety objective will be assessed by:

• Evaluation of any serious adverse device effects upon Sensor insertion through Sensor removal and a follow-up assessment one week (7 ± 3 days) after Sensor removal.

The primary performance objective will be evaluated using the following criteria:

15/20% Performance: Blood glucose measurements from the System must meet the ISO 15197 15/20% accuracy criteria (at least 95% of the matched pairs within ± 15 mg/dL of Comparator values ≤ 75 mg/dL and within ±20% of Comparator values > 75 mg/dL).

DETAILED DESCRIPTION:
Design: Non-randomized, non-treatment, prospective, open label Study.

After providing written informed consent, subjects meeting Inclusion/Exclusion Criteria will be connected to the System for a maximum of 72 hours.

For the purposes of this clinical Study, the System will not display real-time glucose values, glucose trend graphs, or glucose alarms to either the Study Subjects or the Study Site Personnel. There will be no treatment of any Subject based on the output of the System. Diabetes management decisions throughout this Study (if applicable) will be conducted according to hospital procedures.

* 1 set of laboratory measurements will be drawn per Subject for baseline.
* A maximum of 82 blood samples will be drawn per Subject during the 72 hour monitoring session including.

  * Up to 75 blood samples drawn for comparative glucose measurement on laboratory analyzers. Blood samples will be taken from the sampling catheter in the peripheral vein in the contralateral extremity (relative to placement of the System) with no more than 25 samples taken within one day (00:00 to 23:59) for glucose measurement on laboratory analyzers (e.g., Yellow Springs Instrument glucose analyzer (YSI), Radiometer blood analyzer);
  * Up to three (3) sets of laboratory measurements; and
  * Up to 4 other blood samples, as needed. One week (7 + 3 days) after Sensor removal, subjects will be contacted for a follow-up assessment and document any subsequent adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* ICU ≥ 24 hours
* Signed consent

Exclusion Criteria:

* Transplant patient
* Brain injury/surgery patient
* End stage medical conditions or diseases
* Restricted venous access
* History of HIT
* Contraindication for anti-coagulation or bleeding disorder
* Positive pregnancy test
* In other drug, device, or biologic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an anticipated ICU stay of at least 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
15/20% Performance | During 72 hours of anticipated Sensor dwell time
  15/20% Performance: Blood glucose measurements from the System must meet the ISO 15197 15/20% accuracy criteria (at least 95% of the matched pairs within ± 15 mg/dL of Comparator values ≤ 75 mg/dL and within ±20% of Comparator values > 75 mg/dL).

SECONDARY OUTCOMES:
12/12.5% Performance | During 72 hours of anticipated Sensor dwell time
  12/12.5% Performance: Propor-tion of matched pairs meeting within ± 12 mg/dL for Compara-tor values ≤ 100 mg/dL and within ± 12.5% for Comparator values > 100 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Foubert, MD, PhD, Principal Investigator — Onze-Lieve-Vrouwziekenhuis
Locations (2):
- Medical University Graz, Graz, Austria
- Onze-Lieve-Vrouwziekenhuis, Aalst, Belgium